CLINICAL TRIAL: NCT03060070
Title: Comparison of the Analgesic Effect of Ketamine Versus Dexmedetomidine Added to Local Anesthetic in TAP Block for Lower Abdominal Cancer Surgery
Brief Title: Ketamine Versus Dexmedetomidine With Local Anesthetic in TAP Block
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Associte professor, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 321
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Analgesia; Lower Abdominal Cancer
MeSH Terms: interventions — Ketamine; Dexmedetomidine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group, (Placebo Comparator): saline in the same volume will be added to the local anesthetic for TAP block in patients undergoing abdominal cancer surgery
  Interventions: Drug: Ketamine; Drug: dexmedetomidine
- ketamine group, (Active Comparator): ketamine in a dose of 0.5mg/kg will be added to the local anesthetic for TAP block in patients undergoing abdominal cancer surgery
  Interventions: Drug: dexmedetomidine; Drug: control group
- dexmedetomidine group (Active Comparator): dexmedetomidine in a dose of 1ug/kg will be added to the local anesthetic for TAP block in patients undergoing abdominal cancer surgery
  Interventions: Drug: Ketamine; Drug: control group

INTERVENTIONS:
Drug: Ketamine — Ketamine at a dose of 0.5mg/kg will be added to bupivacaine 0.25 (total volume 20ml) in each side using sonar guided TAP block
  Arms: control group,; dexmedetomidine group
Drug: dexmedetomidine — dexmedetomidine at a dose of 1ug/kg will be added to bupivacaine 0.25 (total volume 20ml) in each side using sonar guided TAP block
  Arms: control group,; ketamine group,
Drug: control group — 20ml of 0.25% bupivacaine will be injected in each side of the TAP block
  Arms: dexmedetomidine group; ketamine group,

SUMMARY:
Comparing the analgesic effects of ketamine and dexmedetomidine when added to local anesthetic in TAP block for postoperative analgesia after lower abdominal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients ASA I and II to whom abdominal surgery for cancer will be conducted will be included in the study

Exclusion Criteria:

* Coagulopathies
* ASA III or IV, patient refusal, sensitivity to the used drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative rescue morphine consumption | 24 hours postoperative
  postoperative rescue morphine consumption

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Assiut University, Egypt